CLINICAL TRIAL: NCT05169346
Title: Reducing Neural Perseveration Through Closed Loop Real Time fMRI Neurofeedback to Alleviate Depressive Symptoms
Brief Title: Neurofeedback to Treat Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Yvette Sheline, McLure Professor of Radiology, Neurology and Psychiatry, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 849298; R61MH128492 (NIH)
Record Dates: First submitted 2021-12-08; First posted 2021-12-23 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: MDD

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Neurofeedback (Active Comparator): R61 Phase: Three training sessions. Each training session contains 32 minutes of active neurofeedback runs.
  R33 Phase: Number of training sessions are contingent on R61 findings.
  Interventions: Behavioral: Active Closed Loop Real Time fMRI Neurofeedback
- Sham Neurofeedback (Sham Comparator): R61 Phase: Three training sessions. Each training session contains 32 minutes of sham (placebo) neurofeedback runs.
  R33 Phase: Number of training sessions are contingent on R61 findings.
  Interventions: Behavioral: Sham Closed Loop Real Time fMRI Neurofeedback

INTERVENTIONS:
Behavioral: Active Closed Loop Real Time fMRI Neurofeedback — Active neurofeedback to target neural mechanisms underlying attentional bias in participants with major depressive discover (MDD)
  Arms: Active Neurofeedback
Behavioral: Sham Closed Loop Real Time fMRI Neurofeedback — Sham (placebo) neurofeedback to target neural mechanisms underlying attentional bias in participants with major depressive discover (MDD)
  Arms: Sham Neurofeedback

SUMMARY:
This study tests the efficacy of a new psychotherapeutic strategy for reducing negative attention bias (and therefore depression severity) in participants with MDD (60 in R61 phase and 80 in R33 Phase). This real-time fMRI neurofeedback therapy uses cloud-based pattern classification to decode a patient's attentional state and dynamically modulate task stimuli (in a closed loop) based on this state.

DETAILED DESCRIPTION:
In both the R61and R33 phases we will compare cloud based real time fMRI feedback with placebo (sham feedback) in reducing negative attention bias and depressive symptoms. This study will be the first dose-finding test of real-time fMRI effect on negative attention bias. Measures include: Structured Clinical Interview for DSM-5 (SCID), Clinician-administered diagnostic exam, Montgomery Asberg Depression Rating Scale (MADRS), Clinician-administered scale used to assess the severity of depression, State-Trait Anxiety Inventory (STAI), Self-report questionnaire used to measure types of anxiety and mood symptoms, Mood and Anxiety Symptom Questionnaire (MASQ), Negative perseveration during a go/no-go task, Go/no-go task with overlaid face/scene stimuli; brain response triggers next stimulus, Negative gaze, Negative gaze collected in gaze data following each real time fMRI feedback session

ELIGIBILITY:
Inclusion Criteria:

* gender, inclusive

  * adult aged 18 - 65 meets Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for MDD according to the Clinician-Administered MDD Scale for DSM-5 (unipolar depression or bipolar II depressed)
  * scores at least a minimum score of 16 on Montgomery Asberg Depression Rating Scale (MADRS)
  * normal cognition
  * participants must be able to read and understand English
  * participants must be able to provide consent

Exclusion Criteria:

* pregnancy (female participants)

  * outside age range
  * MRI contraindications (medical implant, claustrophobia, etc.)
  * use of psychoactive medication (including antidepressants) or currently in therapy
  * neurological disorder or any condition that in the view of the PI could impact brain data, cause depression, require medication that could cause depressive symptoms, or otherwise result in participant being unfit for study (for example, co-morbid psychotic, neurological disorders, developmentally or cognitively disabled/impaired, active alcohol or drug abuse/dependence within the past 6 months).
  * non-English speaking
  * non-correctable vision loss
  * refusal to provide informed consent
  * representing an active suicide risk

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Attention Mechanism of Depression | 5 years
  Associate neurofeedback related changes in our hypothesized attentional mechanism of depression (i.e. neural perseveration of negative states) with changes in depression severity as measured by the Montgomery Asberg Depression Rating Scale (MADRS).

CONTACTS AND LOCATIONS:
Overall Officials: Yvette I Sheline, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Neuromodulation in Depression and Stress, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Data will only be shared amongst the study sites.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-04): https://cdn.clinicaltrials.gov/large-docs/46/NCT05169346/Prot_SAP_000.pdf
  • Informed Consent Form (2025-02-18): https://cdn.clinicaltrials.gov/large-docs/46/NCT05169346/ICF_001.pdf